CLINICAL TRIAL: NCT03444350
Title: Evaluating the Clinical and Laboratory Effects of the Use of Ozone in nonsurgıcal perıodontal Treatment : a Randomized Controlled Trial
Brief Title: Use of the Ozone in Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Abubekir Eltas, Director, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inonu University
Record Dates: First submitted 2018-02-14; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Chronic Periodontitis
Keywords: Periodontal treatment; Ozone; oxidative stress
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED TRIAL
Who Masked: Participant, Investigator
Masking Description: The clinician who performed the therapy (S.D.) was not informed about the modality of the treatment till the first session of each patient (right at this moment, a sealed envelope was opened and the clinician was then able to see the treatment modality). The results of the study were evaluated in a blinded manner (both before treatment and after treatment).
  The ozone was applied in the gingival sulcus of all teeth with a fine-tipped tool placed in the periodontal pocket. It was moved in the apical-coronal direction in a sweeping motion. Within 30 seconds, this application was applied in mesial, distal, buccal, and lingual manner. No ozone application was used in the Control Group, and they received only placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (Active Comparator): SRP plus placebo
  Interventions: Device: SRP plus placebo
- Gaseous ozone group (Experimental): SRP plus gaseous ozone [1 W (100 mJ, 10 Hz)]
  Interventions: Device: Gaseous ozone

INTERVENTIONS:
Device: Gaseous ozone — SRP plus gaseous ozone
  Other Names: Ozone DTA
  Arms: Gaseous ozone group
Device: SRP plus placebo — only SRP
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the clinicaland laboratory (as oxidative stress and pro-inflammatory mediators) effects of the use of gaseous ozone in periodontal treatment in addition to scaling and root planning.

The study population consisted of 40 patients with CP (chronic periodontitis). It was performed with two groups; The Test Group, and the Control Group. SRP plus gaseous ozone [1 W (100 mJ, 10 Hz)] was applied to the Test Group. The Control Group, on the other hand, had only SRP.The clinical periodontal parameters were performed and saliva samples were taken before SRP (baseline) and 1 month after treatment. The periodontal examination involved assessing the plaque index, gingival index , probing depth, and clinical attachment level. The total antioxidant status, total oxidant status, nitric oxide, 8-hidroxi-deoksiguanosine, myeloperoxidase, glutathione, malondialdehyde and transforming growth factor-beta levels were determined in the saliva samples.

DETAILED DESCRIPTION:
The study has been designed in a randomized parallelly-controlled and double-blinded design as a full-mouth clinical trial. The duration of the study was 1 month.

The study was performed with two groups; The Test Group, and the Control Group. SRP plus gaseous ozone [1 W (100 mJ, 10 Hz), (n=20)] was applied to the Test Group.

The Control Group, on the other hand, had SRP plus placebo (n=20). The patients were distributed in random order to the 2 groups (each group had 20 patients). One patient in the Ozone Group and 2 patients in the Control Group left the study.

The following clinical periodontal parameters were performed immediately before SRP (baseline), and 1 month after treatment for each test and control groups. Plaque index, GI, PD and CAL were recorded. All clinical parameter measurements were used a manual periodontal probe (PCP- 12, Hu-Friedy, Chicago, IL, USA).

The total antioxidant status, total oxidant status, nitric oxide, 8-hidroxi-deoksiguanosine, myeloperoxidase, glutathione, malondialdehyde and transforming growth factor-beta levels were determined in the saliva samples.

ELIGIBILITY:
Inclusion Criteria:

1. patients having had generalize CP which were agreed upon by consensus at the World Workshop in Periodontics in 1999 [24];
2. three or more teeth having at least two quadrants with probing depth between 4 and 6 mm and radiographic signs of bone loss;
3. aged 30 years and above;
4. a minimum of 20 teeth.

Exclusion Criteria:

1. received periodontal therapy within the last 12 months;
2. systemic diseases which could affect periodontal treatment outcomes;
3. having taken systemic antibiotics within the last 6 months;
4. pregnancy or breast-feeding for female patients.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-05-23 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Laboratory findings | One month
  The total antioxidant status levels ( mmol/L) were determined in the saliva samples.

SECONDARY OUTCOMES:
Clinical findings | One month
  Probing depth was measured the distance between the gingival margin and the deepest aspect of the pocket (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Abubekir Eltas, Ass. Prof., Study Chair — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study has been designed in a randomized parallelly-controlled and double-blinded design as a full-mouth clinical trial. The duration of the study was 1 month. Inonu University Ethics Committee approved the study protocol in accordance with the Helsinki Declaration. Informed Consent Form were received from the participants with their signatures. The participating patients were selected from Inonu University, Department of Periodontology Patient Pool. 40 patients constituted the Study Group.

REFERENCES:
- [Derived] Seydanur Dengizek E, Serkan D, Abubekir E, Aysun Bay K, Onder O, Arife C. Evaluating clinical and laboratory effects of ozone in non-surgical periodontal treatment: a randomized controlled trial. J Appl Oral Sci. 2019 Jan 14;27:e20180108. doi: 10.1590/1678-7757-2018-0108. PMID 30673028